CLINICAL TRIAL: NCT00108160
Title: Intermittent Mupirocin to Prevent Staphylococcal Infection
Brief Title: Preventing Staphylococcal (Staph) Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Michigan (Other); Trinity Health Michigan (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CLNB-001-04S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Staphylococcal Infections
Keywords: mupirocin; prevention and control; s. aureus
MeSH Terms: conditions — Staphylococcal Infections | interventions — Therapeutics; Mupirocin; Polyethylene Glycols; Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mupirocin Ointment [Treatment] (Active Comparator): Treatment arm or active comparator [mupirocin 2% polyethylene glycol (PEG) ointment] will be compared with its placebo comparator [polyethylene glycol (PEF) in patients with a prior history of S. aureus infection. Drug or placebo will be applied topically to nares and/or wounds twice daily for 14 days at 3 month intervals for up to 18 months
  Interventions: Drug: Mupirocin Ointment [Treatment]
- Polyethylene Glycol Ointment [Placebo] (Placebo Comparator): Treatment arm or active comparator [mupirocin 2% polyethylene glycol (PEG) ointment] will be compared with its placebo comparator [polyethylene glycol (PEF) in patients with a prior history of S. aureus infection. Drug or placebo will be applied topically to nares and/or wounds twice daily for 14 days at 3 month intervals for up to 18 months
  Interventions: Drug: Polyethylene Glycol Ointment [Placebo]

INTERVENTIONS:
Drug: Mupirocin Ointment [Treatment] — The impact of the treatment arm versus placebo arm on development of new (recurrent) S. aureus infection will be assessed as the primary end point. Change in S. aureus strains (MSSA versus MRSA) will be assessed as the secondary end point.
  Other Names: Bactroban ointment; Mupirocin 2% in Polyethylene Glycol (PEG) Ointment
  Arms: Mupirocin Ointment [Treatment]
Drug: Polyethylene Glycol Ointment [Placebo] — The impact of the treatment arm versus placebo arm on development of S. aureus re-infections will be assessed as the primary end point. Change in S. aureus strains (MSSA versus MRSA) will be assessed as the secondary end point.
  Other Names: PEG Ointment
  Arms: Polyethylene Glycol Ointment [Placebo]

SUMMARY:
The purpose of this study is to determine if mupirocin 2% in polyethylene glycol (PEG) ointment [Treatment Arm] is effective in preventing moderate to severe re-infection with Staphylococcus aureus compared with treatment with polyethylene glycol (PEG) ointment [Placebo Arm].

DETAILED DESCRIPTION:
Treatment of staphylococcal carriage with the topical antibiotic, mupirocin, has led to decreased infections in some hemodialysis patients and intensive care unit (ICU) patients. However, most of these studies were not placebo controlled and only certain subsets of patients benefited. Relapse of colonization, generally within 90 days after treatment is stopped, presumably with increased risk of infection, approaches 50%. Continuous use of mupirocin on daily, three times weekly, or weekly basis has resulted in increased resistance to the drug. Despite this lack of evidence, the use of mupirocin has become commonplace because it is perceived as an effective and simple means to prevent infection. In a National Institutes on Aging/Claude D. Pepper Older Americans Independence Center (NIA/OAIC)-sponsored proposal, we found that a 2 week treatment regimen with mupirocin ointment was effective in decolonizing older chronically ill nursing home residents of S. aureus when compared with placebo ointment. Decolonization began to decline by 3 months post-treatment, and resistance occurred only once in 52 treated patients. That study was not powered to detect differences in infection between the 2 study groups; the end point was eradication of colonization. However, a trend towards reduction in staphylococcal infection with mupirocin was seen. In addition, there were more therapeutic failures in residents who were colonized with methicillin-resistant S. aureus (MRSA) than methicillin-sensitive S. aureus (MSSA). We hypothesize that intermittent treatment with mupirocin ointment every 3 months may be an effective means of preventing recolonization and infection with S. aureus. We propose to study a patient population that has already had treatment for severe S. aureus infection and is at significant risk for a subsequent infection. Patients will receive mupirocin 2% polyethylene glycol (PEG) ointment [Treatment Arm] or polyethylene glycol (PEG) ointment [Placebo Arm] for 14 days every 3 months. The effect of these two regimens on S. aureus re-infection, re-colonization, and development of mupirocin resistance will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive care at Ann Arbor VA Medical Center, University of Michigan Medical Center, or St. Joseph Mercy Hospital, Ypsilanti who have been hospitalized for documented S. aureus infection will be eligible for enrollment. Staphylococcal infections may be community or hospital-acquired. Patients with S. aureus infection will be identified on a daily basis with the assistance of the Infection Control Practitioner, the Clinical Microbiology Laboratory, the Infectious Diseases Consultation Services, and Infectious Diseases physicians caring for patients in their offices.
* Patients will provide written informed consent. The patient's guardian or next of kin will be contacted for informed consent in the event that the patient is incapable of doing so.

Exclusion Criteria:

* Patients who are unable to cooperate with treatment or follow-up.
* Patients who are not likely to survive beyond one month or those who are transferred back to another acute care hospital.
* Patients who require treatment with rifampin will be excluded since this drug is effective in decolonization of some staphylococcal carriers.
* Patients with known hypersensitivity to mupirocin ointment or polyethylene glycol base.
* Patients with ulcers obviously related to pressure will be excluded because they are frequently large, difficult to keep clean, and infections are difficult to diagnose.
* Patients with small vascular or neuropathic ulcers < 3 cm in circumference and < 2 cm in depth may be enrolled.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2005-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Bradley, MD, Principal Investigator — VA Ann Arbor Healthcare System
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with a history of documented infection with Staphylococcus aureus cared for at Veterans Affairs Ann Arbor Healthcare System, University of Michigan Medical Center, St. Joseph Mercy Hospital (Ypsilanti, MI), and Pittsburgh VA Medical Center from April 2005-August 2012.
Pre-assignment Details: Patients who met study criteria and signed an informed consent were enrolled and randomized to treatment with mupirocin 2% in polyethylene glycol (PEG) ointment or treatment with a placebo (polyethylene glycol) ointment
Groups:
- Mupirocin Ointment (Treatment): Mupirocin 2% in polyethylene glycol (PEG) ointment applied topically to nares and/or wounds for 14 days every 3 months for up to 18 months.
- Polyethylene Glycol Ointment (Placebo): Polyethylene glycol (PEG) ointment applied topically to nares and/or wounds for 14 days every 3 months for up to 18 months.
Period: Overall Study
Arm/Group | Mupirocin Ointment (Treatment) | Polyethylene Glycol Ointment (Placebo)
Started | 83 | 63
Completed Visit 0 (Baseline) | 79 (4 patients who signed consent and were randomized did not complete the initial visit to start drug) | 60 (3 patients who signed a consent and were randomized did not complete the initial visit to start drug)
Completed Visit 1 (2 Wks) | 72 | 54
Completed Visit 2 (3 mo) | 54 | 46
Completed Visit 3 (6 mo) | 44 | 38
Completed Visit 4 (9 mo) | 38 | 37
Completed Visit 5 (12 mo) | 37 | 37
Completed Visit 6 (15 mo) | 36 | 33
Completed Visit 7 (18 mo) | 34 | 31
Completed | 44 (Patients who completed 18 months of mupirocin or developed new (recurrent) S. aureus infection.) | 42 (Participants who completed 18 months of placebo or developed new (recurrent) S. aureus infection.)
Not Completed | 39 | 21
Not completed — Lost to Follow-up | 25 | 12
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Protocol Violation | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Mupirocin Ointment (Treatment): Mupirocin 2% in polyethylene glycol (PEG) ointment applied topically to nares and/or wounds for 14 days every 3 months for up to 18 months (Treatment Group).
- Polyethylene Glycol Ointment (Placebo): Polyethylene glycol (PEG) ointment applied topically to nares and/or wounds for 14 days every 3 months for up to 18 months (Placebo Group).
- Total: Total of all reporting groups
Arm/Group | Mupirocin Ointment (Treatment) | Polyethylene Glycol Ointment (Placebo) | Total
Number analyzed (Participants) | 83 | 63 | 146
Age, Continuous [Mean (Full Range); unit: years] | 56.7 [25 to 88] | 57.9 [22 to 80] | 57.2 [22 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 79 | 54 | 133
Baseline S. aureus Infection Strain [Number; unit: participants]
  MRSA Infection at Baseline | 53 | 43 | 96
  MSSA Infection at Baseline | 30 | 20 | 50

OUTCOME MEASURES:

1. Primary Outcome: Re-infection With S. Aureus
Description: During the study, patients with prior well-documented infections with Staphylococcus aureus who developed new signs and symptoms of infection, met standardized clinical criteria for infection, and had S. aureus isolated on culture were considered to have re-infection with S. aureus. The number of S. aureus re-infections were compared in the mupirocin ointment (Treatment Arm) versus polyethylene glycol ointment (Placebo Arm) for all participants enrolled in the study and in participants who completed each study time point (visit)
Time Frame: 18 months
Population: Re-infections with S. aureus, new or recurrent, were noted for all patients enrolled in the study and for patients who completed each study visit.
Measure: Number; unit: participants with S. aureus re-infection
Arm/Group | Mupirocin Ointment (Treatment) | Polyethylene Glycol Ointment (Placebo)
Number analyzed (Participants) | 83 | 63
participants with S. aureus re-infection
  All enrolled participants [n=83,63)] | 10 | 11
  Completed visit 0 baseline [n=79,60] | 0 | 0
  Completed visit 1 (2 wks) ([n=72,54] | 1 | 0
  Completed visit 2 (3 mo) [n=54,46] | 2 | 3
  completed visit 3 (6 mo) [n=44,38] | 2 | 4
  completed visit 4 (9 mo) [n=38,37] | 3 | 1
  completed visit 5 (12 mo) [n=37,37] | 0 | 0
  completed visit 6 (15 mo) [n=36,33] | 1 | 2
  completed visit 7 (18 mo) [n=34,31] | 1 | 1
Statistical Analysis 1: Comparison: Mupirocin Ointment (Treatment) vs Polyethylene Glycol Ointment (Placebo); Our null hypothesis was that no significant effect of mupirocin ointment (treatment) on S. aureus re-infection would be seen at 18 months compared with placebo ointment. Based on prior studies, we estimated that 198 participants would need to be enrolled assuming a 20% dropout rate; 84 participants per arm would be required to detect a 66% decrease in re-infection from 30% to 10% with a significance level alpha of 0.05 and a power of 0.9; Test type: Superiority or Other; p = 0.356, Chi-squared — No adjustments were made for multiple comparisons

2. Secondary Outcome: Acquisition of New S. Aureus Strains
Description: In the Mupirocin Ointment (Treatment) and Polyethylene Glycol (Placebo) Arms, S. aureus isolates (MSSA or MRSA) that caused infection prior to enrollment in the study were compared with S. aureus infecting isolates (MSSA or MRSA) that occurred during the study (re-infections). Infecting isolates that were found to be MRSA at enrollment and MRSA during the study were considered to be the same strain; this same strain definition was also applied to MSSA isolates. Infecting isolates that changed from MRSA at enrollment to MSSA during the study (or vice versa) were considered to be different strains.
Time Frame: 18 months
Population: Participants with S. aureus re-infection who acquired a new strain during the 18 month study period.
Measure: Number; unit: participants
Arm/Group | Mupirocin Ointment (Treatment) | Polyethylene Glycol Ointment (Placebo)
Number analyzed (Participants) | 10 | 11
participants
  Same strain baseline & Re-infection | 10 | 10
  MRSA Baseline & Re-Infection | 8 | 10
  MSSA Baseline & Re-Infection | 2 | 0

3. Other Pre Specified Outcome: S. Aureus Re-infections (New or Recurrent)
Description: The anatomic site of each S. infection at enrollment and S. aureus re-infection that occurred during the study was compared. S. aureus isolated from a different site of infection than at baseline was considered to represent a new infection. Isolation of S. aureus from the same site as the baseline infection was considered to represent a recurrent infection.
Time Frame: 18 months
Measure: Number; unit: participants
Groups:
- Mupirocin Ointment [Treatment]: Mupirocin 2% in polyethylene glycol (PEG) ointment applied topically to nares and/or wounds for 14 days every 3 months for up to 18 months.
- Polyethylene Glycol Ointment [Placebo]: Polyethylene glycol (PEG) ointment applied topically to nares and/or wounds for 14 days every 3 months for up to 18 months.
Arm/Group | Mupirocin Ointment [Treatment] | Polyethylene Glycol Ointment [Placebo]
Number analyzed (Participants) | 10 | 11
participants
  All Re-Infections | 10 | 11
  Re-infections Different Anatomic Site | 7 | 6

ADVERSE EVENTS:
Time Frame: Duration of the study - 18 months
Description: A questionnaire was administered by study personnel at each visit. Patients who did not show for visits were contacted by phone and mail at regular intervals by study personnel. Chart reviews were conducted for patients who did not show or respond.
Groups:
- Mupirocin Ointment: Mupirocin 2% in polyethylene glycol (PEG) ointment applied topically to nares and/or wounds for 14 days every 3 months for up to 18 months.
- Polyethylene Glycol Ointment: Polyethylene glycol (PEG) ointment applied topically to nares and/or wounds for 14 days every 3 months for up to 18 months.
Arm/Group | Mupirocin Ointment | Polyethylene Glycol Ointment
Serious Adverse Events (participants affected / at risk) | 1/83 | 2/63
Other Adverse Events (participants affected / at risk) | 0/83 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mupirocin Ointment (N=83) | Polyethylene Glycol Ointment (N=63)
Underlying condition that led to death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — breast cancer metastatic
Underlying condition that led to death (Cardiac disorders) | 1 (1) | 1 (1) — Congestive heart failure

LIMITATIONS AND CAVEATS:
The study is underpowered to detect differences between the two treatment arms. We achieved only 75% of target enrollment, and 41.1% dropped out before reaching a primary endpoint. Our re-infection rate was also lower than anticipated (14.4%).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No